CLINICAL TRIAL: NCT01608386
Title: Anterior Approach Combined With Infrahepatic Inferior Vena Cava Clamping Right Hepatic Resection for Large Hepatocellular Carcinoma: A Prospective Randomized Controlled Study
Brief Title: A Study of Anterior Approach Combined With Infrahepatic Inferior Vena Cava Clamping
Acronym: AA+IVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Chengjun Sui,MD, Clinical Professor, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2012-002-16
Record Dates: First submitted 2012-05-22; First posted 2012-05-31 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Surgical Approach & Incisions; Blood Loss
Keywords: Anterior approach; infrahepatic inferior vena cava clamping; hepatic resection
MeSH Terms: conditions — Surgical Wound; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anterior approach+IVC clamping (Experimental): Use anterior approach combined with infrahepatic Inferior Vena Cava clamping in right hepatectomy for HCC patients.
  Interventions: Procedure: IVC clamping
- anterior approach (No Intervention): Only use anterior approach in right hepatectomy for HCC patients.

INTERVENTIONS:
Procedure: IVC clamping — in right hepatectomy,use anterior approach and infrahepatic Inferior Vena Cava clamping.
  Arms: anterior approach+IVC clamping

SUMMARY:
Anterior approach results in better operative and survival outcomes compared with the conventional approach in patients with large hepatocellular carcinoma (HCC), but anterior approach has the problem of bleeding from the hepatic vein.

Our previous study showed that infrahepatic inferior vena cava (IVC) clamping can reduce blood loss during conventional hepatic resection. The investigators guess infrahepatic IVC clamping may also reduce blood loss in anterior approach right hepatic resection. So the investigators conduct this prospective, randomized, controlled trial to compare anterior approach combined with infrahepatic IVC clamping and anterior approach in major right hepatectomy for large HCC.

DETAILED DESCRIPTION:
Traditionally, mobilisation of the right hemiliver followed by right hepatic vein control before parenchymal transection has been considered the standard approach to a major right hepatectomy. However, this approach is often difficult and hazardous when performing liver resection for large hepatocellular carcinoma (HCC) or for tumors with extrahepatic organ invasion in the right retrohepatic region.In setting of right hepatectomy by an anterior approach,liver mobilisation is performed only at the end of parenchymal transection, when all vascular connections have already been interrupted.The anterior approach was found to be associated with significantly less intraoperative blood loss, less blood transfusions and a lower hospital mortality rate.However,excessive bleeding can occur at the deeper plane of parenchymal transection from the right hepatic vein or middle hepatic vein.

Bleeding from the hepatic veins is closely related to the CVP.Our previous retrospective analysisfound that the infrahepatic inferior vena cava (IVC) clamping is efficacious in reducing CVP without the need of systemic fluid restriction and is associated with significantly less intraoperative blood loss during complex hepatectomy.

The aim of the present study was therefore to evaluate if the application of the anterior approach combined with infrahepatic IVC clamping during right hepatectomy for large HCC reduces intraoperative blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and being willing to sign the informed consent form
* Aged 18-75 years
* Diagnosed HCC by clinical findings and radiography，tumor size ≥ 5cm and located in the right lobe, need to perform right hemihepatectomy or major right hepatic resection (three Couinaud's segments)
* Without any surgery contraindication
* Child-Pugh grade A

Exclusion Criteria:

* Refusal to take part in the study
* With lymph node or extrahepatic metastases
* History of previous hepatectomy or other abdominal operation
* Those who can not be follow-up
* Non-HCC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
intraoperative total blood loss | participants will be followed for the duration of the entire operation,an expected average of 140 minutes

SECONDARY OUTCOMES:
operation time | the duration of the entire operation,an expected average of 140 minutes
intraoperative CVP value | participants will be followed for the duration of the parenchymal transection,an expected average of 20 minutes
morbidity and mortality | participants will be followed for the duration of the postoperative hospital stay,an expected average of 15 days
postoperative hepatorenal function | postoperative day 1,3 and 7
postoperative hospital stay | the duration of the postoperative hospital stay,an expected average of 15 days
disease-free survival duration and overall survival duration | the duration from operation to recurrence or death,an expected average of 3 years
blood loss during parenchymal transection | the duration of the parenchymal transection,an expected average of 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jiamei Yang, MD, Study Director — Eastern Hepatobiliary Surgery Hospital; Chengjun Sui, MD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital